CLINICAL TRIAL: NCT04984733
Title: An Open Label Single Arm Phase II Trial in Patients With Advanced Unresectable Previously Treated Oesophagogastric Adenocarcinoma Which is MGMT Deficient
Brief Title: Temozolomide + Nivolumab in MGMT Methylated Oesophagogastric Cancer
Acronym: ELEVATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 61191
Record Dates: First submitted 2021-01-13; First posted 2021-07-30 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Adenocarcinoma - GEJ; Cancer of Esophagus
Keywords: cancer; Oesophagogastric; Oesophagogastric adenocarcinoma,; MGMT deficient,; O6-methylguanine-DNA-methyltransferase; MGMT protein, human; MGMT methylated
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms | interventions — Temozolomide; Nivolumab

STUDY DESIGN:
Intervention Model Description: An open-label, single arm, A'Hern single stage phase II design. Patients will receive TMZ priming followed by nivolumab to establish disease control rates.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Metronomic TMZ 50mg/m2/day orally for 3 months, then nivolumab 240mg IV until progression.
  Metronomic TMZ 50mg/m2/day orally until progression then nivolumab 240mg IV until progression. Patients who progress on TMZ will start monotherapy with nivolumab.
  Metronomic TMZ50mg/m2/day orally for 3 months, then nivolumab 240mg IV +/- TMZ until progression. Patients who don't progress on TMZ will commence with combination treatment; TMZ + Nivolumab at 3 mths until they progress
  Metronomic TMZ 50mg/m2/day orally for 3 months, then nivolumab 240mg IV +/- TMZ until 24 months. Patients will remain on combination therapy up to a maximum of 24mths.
  Interventions: Drug: Temozolomide; Drug: Temozolomide 50mg/m2/day; Drug: Temozolomide 3 month; Drug: Temozolomide 24month

INTERVENTIONS:
Drug: Temozolomide — Metronomic TMZ 50mg/m2/day orally for 3 months then nivolumab 240mg IV +/- TMZ until progression.
  Patients who don't progress on TMZ will commence with combination treatment; TMZ + Nivolumab at 3 mths. Patients who progress on TMZ will start monotherapy with nivolumab. Patients will remain on monotherapy with nivolumab or combination therapy until progression or up to a maximum of 24mths.
  Other Names: Nivolumab
Drug: Temozolomide 50mg/m2/day — Metronomic TMZ 50mg/m2/day orally until progression then nivolumab 240mg IV until progression
  Other Names: Nivolumab
Drug: Temozolomide 3 month — Metronomic TMZ 50mg/m2/day orally for 3 months, then nivolumab 240mg IV and TMZ until progression.
  Other Names: Nivolumab
Drug: Temozolomide 24month — Metronomic TMZ 50mg/m2/day orally for 3 months, then nivolumab 240mg IV and TMZ until a maximum of 24 months
  Other Names: Nivolumab

SUMMARY:
An open label single arm phase II trial in patients with advanced unresectable previously treated oesophagogastric adenocarcinoma which is MGMT deficient.

DETAILED DESCRIPTION:
The aim of the ELEVATE trial is to determine the activity and safety of maintenance TMZ dosing followed by nivolumab treatment to evaluate the potential for a future randomised trial against a standard of care control arm. The rationale to continue TMZ for 3 months or until PD is to evaluate the emergence of mismatch repair deficiency both with and without radiological PD, as clinically relevant MMRd may emerge before radiological progression. This will also reduce the number of patients who drop out due to symptomatic progressive disease.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients ≥ 18 years of age
* Pathologically confirmed advanced unresectable or metastatic OGA
* MGMT methylation on archival tissue
* Mismatch repair proficient (MSI-normal or MMR intact)
* Previously treated with at least 3 months of platinum and fluoropyrimidine based chemotherapy for advanced disease and without evidence of disease progression.
* Measurable disease per RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Can swallow TMZ capsules
* Adequate organ function assessed within 7 days before randomization:

  * White blood cell count (WBC) > 1.5 x 109/L
  * Absolute neutrophil count (ANC) > 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Haemoglobin ≥ 90 g/L
  * Measured/calculated creatinine clearance ≥ 60 mL/min (according to Cockroft-Gault formula).
  * Total bilirubin within normal limits (if the patient has documented Gilbert's disease ≤ 1.5 x ULN or direct bilirubin ≤ 1.5 x ULN)
  * Aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 1.5 x ULN
* All toxicities (exception alopecia, and grade 2 fatigue, neuropathy and lack of appetite /nausea) attributed to prior anti-cancer therapy must have resolved to grade 1 (NCI CTCAE version 5.0) or baseline before administration of study drug.
* Women of childbearing potential (WOCBP) may be included following a confirmed menstrual period and must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG)). Pregnancy test must be within 24 hours prior to starting treatment. (A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient).
* WOCBP should use one highly effective and one effective method of birth control during the study treatment period and for at least 5 months after the last dose of the study treatment.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 5 months after the last dose of the study treatment.
* Men who are sexually active with a WOCBP must adhere to contraception during and for a period of 7 months after the last dose of the study treatment.
* Absence of any psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Written informed consent

EXCLUSION CRITERIA

* Previous treatment with TMZ
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Active central nervous system metastases
* Candidate for curative surgery
* Previous malignancies are excluded unless a complete remission was achieved at least 5 years prior to study entry. Adequately treated cervical carcinoma in situ, and localized non-melanoma skin cancer are not exclusion criteria, regardless of timepoint of diagnosis.
* Active, known, or suspected infectious or autoimmune disease (except for patients with Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enrol)
* Conditions requiring systemic treatment with either corticosteroids (≥ 10 mg daily prednisolone or equivalent) or other immunosuppressive medications within 14 days of study drug administration
* Interstitial lung disease
* > Grade 1 peripheral neuropathy
* Positive test result for HBV or HCV indicating acute or chronic infection
* Known history of testing positive for HIV or known AIDS
* Known hypersensitivity to the components or excipients of co-trimoxazole, temozolomide or nivolumab. (Please refer to nivolumab IB and SmPC for TMZ and co-trimoxazole).
* Known hypersensitivity to dacarbazine (DTIC)
* Clinically significant abnormal 12-lead ECG. If clinically indicated, cardiac function assessment using either echocardiography or MUGA Scan, if clinically significant the patient is ineligible.
* In the past 6 months serious cardiac illness or medical condition including but not confined to:

  * History of documented congestive heart failure (CHF)
  * High-risk uncontrolled arrhythmias
  * Angina pectoris requiring antianginal medication
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction
  * Poorly controlled hypertension (e.g. systolic >180mm Hg or diastolic greater than 100mm Hg)
* Patients with severe liver parenchymal damage
* Patients with severe renal insufficiency where repeated measurements of the plasma concentration cannot be performed
* Patients with a history of drug-induced immune thrombocytopenia with use of trimethoprim and/or sulfonamides.
* Patients with acute porphyria
* Patients with severe myelosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Tumour Response to nivolumab | 24 months
  To determine the anti-tumour activity of nivolumab, when given after temozolomide in patients with previously treated advanced oesophagogastric adenocarcinoma which are MGMT methylated.

SECONDARY OUTCOMES:
The percentage of patients who have achieved response | 6 months
  The Disease control rate determine the effect of TMZ priming followed by nivolumab on disease control rates of patients with previously treated advanced oesophagogastric adenocarcinoma which is MGMT methylated.
  Disease control rate, according to RECIST v1.1 and iRECIST, 6 months after starting nivolumab, and 3 months after starting TMZ, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Smyth, Principal Investigator — Cambridge University
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No